CLINICAL TRIAL: NCT06565468
Title: The Effect of Cold Water Immersion on Recovery and Performance in NCAA Division I Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Collaborators: Whoop Inc. (Industry)
Responsible Party: Principal Investigator, Joshua T. Goldman, MD, MBA, Associate Professor in the Departments of Family Medicine and Orthopaedic Surgery, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: UCLACWI
Record Dates: First submitted 2024-08-16; First posted 2024-08-22 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Recovery, Physiological; Athletic Performance

STUDY DESIGN:
Intervention Model Description: Cohort cross-over design. The study population will be randomized into two cohorts. The first cohort will begin with the control phase and then transition to the intervention phase. The second cohort will begin with the intervention phase and then transition to the control phase.
Masking Description: Collected data will be stored and managed using REDCap secure web-based database management system. Any personally identifiable information will be coded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Cold water immersion phase. (Experimental)
  Interventions: Device: Cold water immersion pool.
- Control phase. (No Intervention)

INTERVENTIONS:
Device: Cold water immersion pool. — Participants will complete a session of cold-water immersion within one hour of finishing the last training session of the day. Cold water immersion will consist of ten minutes of submersion to the neck in a cold-water tub with a target temperature of 55 degrees Fahrenheit (daily temperatures will be recorded at the time of each session). The acceptable range for the cold water immersion protocol will be from 53-57 degrees Fahrenheit. The immersion process will not be completed if the temperature of the water is outside of this range. Participants will complete five sessions per week, with a total of 10 sessions to be completed over the 14-day intervention.
  Arms: Cold water immersion phase.

SUMMARY:
In this study, the investigators will examine the effect of cold-water immersion (CWI) on objective and subjective recovery metrics, as well as simple performance metrics, in National Collegiate Athletics Association (NCAA) Division I Men's and Women's Volleyball players, Men's Football players, and Men's and Women's Cross Country runners. This is a cohort cross-over study that will take place over the course of four weeks during an intensive training cycle. Participants will wear a WHOOP monitoring device on their wrists at all times during the study period. The two-week intervention will consist of ten minutes of CWI to take place within one hour of the completion of the last training session of the day. The target water temperature will be 55 degrees Fahrenheit, and each participant will complete five sessions of CWI per week (for a total of ten sessions over the two-week intervention phase). Objective recovery measures will include heart rate variability, resting heart rate, total sleep time, slow wave sleep time, sleep consistency, blood oxygenation, and nocturnal skin temperature, all of which will be collected continuously by the WHOOP monitoring device. Subjective recovery measures will include three surveys to be completed daily, including the Likert Scale of Muscle Soreness, the Total Quality Recovery Scale, and the Single-Item Sleep Questionnaire. Performance measures will include a counter-movement jump to be completed two times per week, an isometric mid-thigh pull to be completed once per week, and a drop jump to be completed once per week. These outcome measures will similarly be collected during the two-week control period, during which participants will not have access to CWI following training sessions.

DETAILED DESCRIPTION:
This is a cohort cross-over design that will take place over four weeks during an intensive training cycle. The study population will be randomized into two cohorts. The first cohort will begin with the control phase and then transition to the intervention phase. The second cohort will begin with the intervention phase and then transition to the control phase.

Control phase:

Participants will complete normal training sessions over a 14-day period and will not have access to cold water immersion (CWI) during this time.

Intervention phase:

Participants will complete normal training sessions over a 14-day period. They will complete a session of CWI within one hour of finishing the last training session of the day. CWI will consist of ten minutes of submersion to the neck in a cold-water tub with a target temperature of 55 degrees Fahrenheit (daily temperatures will be recorded at the time of each session). The acceptable range for the CWI protocol will be from 53-57 degrees Fahrenheit. The immersion process will not be completed if the temperature of the water is outside of this range. Participants will complete five sessions per week, with a total of 10 sessions to be completed over the 14-day intervention.

Participants will wear a WHOOP 4.0 wrist device throughout the entire four-week study period to collect continuous biometric data and to monitor sleep patterns overnight. Athletic performance testing will consist of a counter-movement jump completed two times per week, an isometric mid-thigh pull completed one time per week, and a drop jump completed one time per week. Participants will complete three surveys daily over the four-week period. Participants will be aware of their performance testing metrics and physiologic measures as reported in the WHOOP app.

Physiological Measures:

Biometric Monitoring:

Participants will be asked to wear a WHOOP 4.0 wrist device throughout the entirety of the study period. This device will provide continuous biometric data including resting heart rate, exertional heart rate, heart rate variability, respiratory rate, blood oxygenation, and skin temperature.

Sleep Monitoring:

Participants will be asked to wear a WHOOP 4.0 wrist device throughout the entirety of the study period, which will provide detailed data regarding sleep quantity, quality, consistency, and efficiency. It will also provide information about the time spent in each phase of sleep (light, REM, slow wave [deep], and awake) and respiratory rate throughout sleep.

Athletic Performance Testing:

Counter-movement jump:

The Counter-movement Jump (CMJ) is a vertical jump test performed by having an athlete quickly squat on a force plate to a self-selected depth and then jump as high as possible. It is primarily used for monitoring sports performance, inter-limb asymmetries, neuromuscular fatigue, and the effectiveness of different training programs.

Isometric mid-thigh pull:

The Isometric Mid-Thigh Pull (IMTP) is performed on a dual force plate system with a barbell locked at mid-thigh height, with the athlete attempting to produce as much force as possible as quickly as possible. The test requires an individual to pull on a fixed barbell while standing on the force plate system with a maximal effort for 3-5 seconds. It has been used in studies that evaluated the effects of resistance training programs on maximum strength development, the acute ergogenic effects of supplements on strength (e.g., sodium bicarbonate, caffeine), and the influence of motor learning strategies on maximum force production. Additionally, the isometric mid-thigh pull test is also used to assess fatigue and recovery from exercise and competition.

Drop jump:

The drop jump is a fitness test of leg strength and power which requires the athlete to "drop off" a box and immediately jump as high as they can. The athlete stands on a box, adjacent to the force plate. The athlete then drops down off the box onto the force plate, bending the knees on landing, then immediately performs a maximal vertical jump. The athlete jumps vertically as high as possible, and lands back on the mat with both feet landing at the same time. This test is designed to assess average power and reactive strength.

Perceptual Measure and Questionnaires:

Single-Item Sleep Quality Scale (SISQ):

Participants will be asked to complete the single-item sleep quality scale daily. This survey has been validated against the Pittsburgh Sleep Quality Index (PSQI) for assessment of subjective sleep quality. Participants will rate the quality of their sleep on a scale of 1-10. The survey will consist of the following prompt: "Please think about the quality of the participant's sleep overall, such as how many hours of sleep the participant got, how easily the participant fell asleep, how often the participant woke up during the night (except to go to the bathroom), how often the participant woke up earlier than the participant had to in the morning, and how refreshing the participant's sleep was. Over the past seven days, how would the participant rate the participant's sleep quality overall? (Mark only one box from 0-10, with 0 being terrible, 1-3 being poor, 4-6 being fair, 7-9 being good, and 10 being excellent)."

Total Quality Recovery Scale (TQR):

Participants will be asked to complete this survey daily. This tool is an overall measure of perception of recovery on a 6-20 point scale, estimating the perception of recovery daily to detect the current form of athletes and to monitor short-lived emotional changes. The TQR scale is similar to the perceived exertion scale and is used as a means to measure psycho-physiological recovery. A score for the TQR is ideal at a value of 20, and a score of 13 is considered the minimum score; any scores below this indicate that recovery is incomplete.

Likert Scale of Muscle Soreness (LSMS):

Participants will be asked to complete this survey daily. This tool is a measure of lower limb muscle soreness and has been validated against the Visual Analog Scale in athletes. The survey assesses subjective ratings of lower body soreness (quadriceps, hamstrings) ranging from 0-6 (0 = complete absence of pain; 1 = light pain felt only when touched/a vague ache; 2 = moderate pain felt only when touched/a slight persistent pain; 3 = light pain when walking up or down stairs; 4 = light pain when walking on a flat surface/painful; 5 = moderate pain, stiffness, or weakness when walking/very painful; and 6 = severe pain that limits my ability to move).

Medical Equipment:

In-ground Cold Plunge Pool:

The investigators will be utilizing the in-ground cold plunge pools located in the UCLA athletic training rooms. The water in the pool is chlorinated and checked and maintained at a 1.0-1.2 ppm by a CPO (certified pool operator) daily. There is a recirculating sand/silicate filtration system. All study participants will be required to shower prior to use and follow all Occupational Safety and Health Administration (OsHA protocols, in line with the Campus Department of Health and Safety. Additionally, the pools have a UV sanitization system. There are grab rails on all steps/stairs, as well as non-skid grips on steps to reduce the risk of slips and falls.

ELIGIBILITY:
Inclusion Criteria:

* Male and female student-athletes aged 18 years or older
* Currently enrolled at UCLA and participating in the following National Collegiate Athletics Association (NCAA) Varsity sports: Men's and Women's Volleyball, Football, Men's and Women's Cross Country.

Exclusion Criteria:

* Must meet above inclusion criteria.
* Unable to complete the required physical testing due to injury or other impairment.
* Age less than 18 years old at time of enrollemnt
* Open wounds or broken skin
* History of hypersensitivity to cold, including but not limited to Raynaud's phenomenon, cold urticaria, cryoglobulinemia, and paroxysmal cold hemoglobinuria
* Under the influence of drugs or alcohol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Heart-rate variability | Four week time period
  As measured by WHOOP 4.0 wrist device

SECONDARY OUTCOMES:
Resting heart rate | Four week time period
  As measured by WHOOP 4.0 wrist device
Total Sleep Time | Four week time period
  As measured by WHOOP 4.0 wrist device
Slow Wave Sleep Time | Four week time period
  As measured by WHOOP 4.0 wrist device
Sleep Consistency | Four week time period
  As measured by WHOOP 4.0 wrist device
Blood Oxygenation | Four week time period
  As measured by WHOOP 4.0 wrist device
Nocturnal Skin Temperature | Four week time period
  As measured by WHOOP 4.0 wrist device
Likert Scale of Muscle Soreness | Four week time period
  Survey
Total Quality Recovery Scale | Four week time period
  Survey
Single Item Sleep Questionnaire | Four week time period
  Survey
Counter Movement Jump | Four week time period
  Performance Metric
Isometric Mid-Thigh Pull | Four week time period
  Performance Metric
Drop Jump | Four week time period
  Performance Metric

CONTACTS AND LOCATIONS:
Locations (1):
- UCLA Orthopedics, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ravier G, Marcel-Millet P, Fostel C, Baradat E. Post-Exercise Cold- and Contrasting-Water Immersion Effects on Heart Rate Variability Recovery in International Handball Female Players. J Hum Kinet. 2022 Feb 10;81:109-122. doi: 10.2478/hukin-2022-0010. eCollection 2022 Jan. PMID 35291638
- [Background] Laborde S, Wanders J, Mosley E, Javelle F. Influence of physical post-exercise recovery techniques on vagally-mediated heart rate variability: A systematic review and meta-analysis. Clin Physiol Funct Imaging. 2024 Jan;44(1):14-35. doi: 10.1111/cpf.12855. Epub 2023 Oct 2. PMID 37754676
- [Background] Moore E, Fuller JT, Buckley JD, Saunders S, Halson SL, Broatch JR, Bellenger CR. Impact of Cold-Water Immersion Compared with Passive Recovery Following a Single Bout of Strenuous Exercise on Athletic Performance in Physically Active Participants: A Systematic Review with Meta-analysis and Meta-regression. Sports Med. 2022 Jul;52(7):1667-1688. doi: 10.1007/s40279-022-01644-9. Epub 2022 Feb 14. PMID 35157264
- [Background] Poignard M, Guilhem G, Jubeau M, Martin E, Giol T, Montalvan B, Bieuzen F. Cold-water immersion and whole-body cryotherapy attenuate muscle soreness during 3 days of match-like tennis protocol. Eur J Appl Physiol. 2023 Sep;123(9):1895-1909. doi: 10.1007/s00421-023-05190-8. Epub 2023 Apr 23. PMID 37088821
- [Background] Seco-Calvo J, Mielgo-Ayuso J, Calvo-Lobo C, Cordova A. Cold Water Immersion as a Strategy for Muscle Recovery in Professional Basketball Players During the Competitive Season. J Sport Rehabil. 2020 Mar 1;29(3):301-309. doi: 10.1123/jsr.2018-0301. PMID 30676280
- [Background] Roberts LA, Raastad T, Markworth JF, Figueiredo VC, Egner IM, Shield A, Cameron-Smith D, Coombes JS, Peake JM. Post-exercise cold water immersion attenuates acute anabolic signalling and long-term adaptations in muscle to strength training. J Physiol. 2015 Sep 15;593(18):4285-301. doi: 10.1113/JP270570. Epub 2015 Aug 13. PMID 26174323
- [Background] Grgic J. Effects of post-exercise cold-water immersion on resistance training-induced gains in muscular strength: a meta-analysis. Eur J Sport Sci. 2023 Mar;23(3):372-380. doi: 10.1080/17461391.2022.2033851. Epub 2022 Feb 20. PMID 35068365
- [Background] Haq A, Ribbans WJ, Hohenauer E, Baross AW. The Comparative Effect of Different Timings of Whole Body Cryotherapy Treatment With Cold Water Immersion for Post-Exercise Recovery. Front Sports Act Living. 2022 Jul 6;4:940516. doi: 10.3389/fspor.2022.940516. eCollection 2022. PMID 35873209
- [Background] Moore E, Fuller JT, Bellenger CR, Saunders S, Halson SL, Broatch JR, Buckley JD. Effects of Cold-Water Immersion Compared with Other Recovery Modalities on Athletic Performance Following Acute Strenuous Exercise in Physically Active Participants: A Systematic Review, Meta-Analysis, and Meta-Regression. Sports Med. 2023 Mar;53(3):687-705. doi: 10.1007/s40279-022-01800-1. Epub 2022 Dec 17. PMID 36527593
- [Background] Garcia CA, da Mota GR, Marocolo M. Cold Water Immersion is Acutely Detrimental but Increases Performance Post-12 h in Rugby Players. Int J Sports Med. 2016 Jul;37(8):619-24. doi: 10.1055/s-0035-1565200. Epub 2016 May 2. PMID 27136509
- [Background] Al Haddad H, Parouty J, Buchheit M. Effect of daily cold water immersion on heart rate variability and subjective ratings of well-being in highly trained swimmers. Int J Sports Physiol Perform. 2012 Mar;7(1):33-8. doi: 10.1123/ijspp.7.1.33. Epub 2011 Aug 30. PMID 21941017
- [Background] Anicic Z, Janicijevic D, Knezevic OM, Garcia-Ramos A, Petrovic MR, Cabarkapa D, Mirkov DM. Assessment of Countermovement Jump: What Should We Report? Life (Basel). 2023 Jan 9;13(1):190. doi: 10.3390/life13010190. PMID 36676138
- [Background] Grgic J, Scapec B, Mikulic P, Pedisic Z. Test-retest reliability of isometric mid-thigh pull maximum strength assessment: a systematic review. Biol Sport. 2022 Mar;39(2):407-414. doi: 10.5114/biolsport.2022.106149. Epub 2021 Jun 1. PMID 35309521
- [Background] Tong Z, Chen W, Xu H, Zhai F. Optimal Loading Height: A Practical Research of Drop Jump from Biomechanics. J Healthc Eng. 2022 Mar 15;2022:4173639. doi: 10.1155/2022/4173639. eCollection 2022. PMID 35340227
- [Background] Snyder E, Cai B, DeMuro C, Morrison MF, Ball W. A New Single-Item Sleep Quality Scale: Results of Psychometric Evaluation in Patients With Chronic Primary Insomnia and Depression. J Clin Sleep Med. 2018 Nov 15;14(11):1849-1857. doi: 10.5664/jcsm.7478. PMID 30373688
- [Background] Selmi O, Ouergui I, Muscella A, My G, Marsigliante S, Nobari H, Suzuki K, Bouassida A. Monitoring Psychometric States of Recovery to Improve Performance in Soccer Players: A Brief Review. Int J Environ Res Public Health. 2022 Jul 31;19(15):9385. doi: 10.3390/ijerph19159385. PMID 35954741
- [Background] Impellizzeri FM, Maffiuletti NA. Convergent evidence for construct validity of a 7-point likert scale of lower limb muscle soreness. Clin J Sport Med. 2007 Nov;17(6):494-6. doi: 10.1097/JSM.0b013e31815aed57. PMID 17993794